CLINICAL TRIAL: NCT07123194
Title: The Effect of Art-Based Nursing Intervention Helping to Develop Healthy Digital Habits on Digital Addiction, Cyberbullying and Self-Efficacy in Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Esra Unal, Research Assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUnal202575
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Digital Addiction; Art Therapy; Cyberbullying; Self Efficacy; Adolescence
Keywords: Art Therapy; Digital Addiction; Cyberbullying; Self-Efficacy; Adolescent
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Intervention Model Description: This research is an experimental type, randomized controlled study designed in a pre-test post-test design.
Masking Description: Statistician and language translator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arts-Based Nursing Intervention Program (Experimental): An 8-week "Art-Based Nursing Intervention Program to Help Gain Healthy Digital Habits" will be implemented.
  Interventions: Behavioral: An Arts-Based Nursing Intervention Program to Help Develop Healthy Digital Habits
- Usual School Schedule (Control) (No Intervention): No intervention will be applied to the control group. However, after the experimental group completes its interventions, the "Arts-Based Nursing Intervention Program to Help Develop Healthy Digital Habits" will be applied to the control group at a timeframe deemed appropriate by school administrators and in a manner that will not disrupt students' classes.

INTERVENTIONS:
Behavioral: An Arts-Based Nursing Intervention Program to Help Develop Healthy Digital Habits — Session Time: Arts-Based Nursing Intervention Program Sessions to Help Develop Healthy Digital Habits Week 1, Session 1 - Introductions and Group Agreement Formation (60 minutes) Week 2, Session 2 - Where Am I in the Digital World? (60 minutes) Week 3, Session 3 - Digital Addiction: Are You Connected or Addicted? (90 minutes) Week 4, Session 4 - Digital Addiction and Its Effects (90 minutes) Week 5, Session 5 - Digital Danger: Cyberbullying (90 minutes) Week 6, Session 6 - Discovering Strengths: The Relationship Between Digital Addiction and Self-Efficacy (90 minutes) Week 7, Session 7 - Digital Detox and Alternatives (90 minutes) Week 8, Session 8 - Evaluation and Closing (90 minutes)
  Arms: Arts-Based Nursing Intervention Program

SUMMARY:
In today's world where digital technologies are integrated into every aspect of life, adolescents' unhealthy and uncontrolled use of digital media causes important psychosocial problems such as digital addiction and cyberbullying. This research aims to examine the effects of an art-based nursing intervention program in order to help adolescents born into the digital world gain healthy digital habits. The art-based nursing intervention program that helps gain healthy digital habits aims to increase adolescents' expressive expression skills, develop their skills in coping with challenging situations in the digital environment and strengthen their self-efficacy levels through creative art activities. The research is a randomized controlled trial designed as an experimental type, pre-test-post-test design. The research will be carried out in Prof. Dr. Fuat Sezgin Secondary School in Karatay district of Konya province. The sample group was determined as a total of 64 adolescents, 32 intervention and 32 control. Adolescents will be randomly assigned to the intervention and control groups. The pre-test data of the intervention and control groups were collected before the program started; The post-test data will be collected face-to-face by the researcher after the program is completed using the Personal Information Form, Digital Addiction Scale for Children, Revised Cyberbullying Scale (YSZE-II) and Self-Efficacy Scale for Children. It is expected that the digital addiction and cyberbullying levels of adolescents who are applied the art-based nursing intervention program that helps them gain healthy digital habits will be lower than the control group, and their self-efficacy levels will be higher than the control group. It is anticipated that the findings to be obtained as a result of the research will enable the development of creative and holistic intervention approaches that will increase the functionality of school health nurses against the risks posed by the digital age on young people. It is also thought that it can provide an evidence-based basis for the usability of art-based interdisciplinary practices in the field.

DETAILED DESCRIPTION:
The rapid development of twenty-first-century technology and the integration of digital devices such as smartphones, tablets, laptops, or desktop computers into daily life are leading to radical changes in individuals' lifestyles, and this has brought to the fore the concept of digital addiction, which is considered a significant public health problem. Digital addiction is not yet included in an official psychiatric diagnostic category according to the DSM-V or DSM-IV TR. However, within the relevant literature, digital addiction is defined as the compulsive and uncontrolled use of technological devices and is therefore considered under the umbrella of behavioral addictions. Furthermore, it has been noted that, just like behavioral addictions, digital addiction causes various psychosocial problems in the individual. In this context, nursing interventions aimed at reducing the risk of digital addiction and strengthening public mental health are considered to be of increasing importance. The new world order is making technology a necessity, not a choice, for individuals. It is also noted that familiarity with digital tools is a significant factor influencing digital addiction. In this regard, it is frequently stated in many studies on the subject that adolescents, born in an era when digital tools are widely used, who can use technological devices with natural competence and are referred to as "digital natives," are a vulnerable group for digital addiction. For example, according to the Turkish Statistical Institute's Children's Information Technology Use Survey, 91.3% of children aged 6-15 actively use the internet, and 76.1% of this age group own a personal mobile phone. The same study also reports that the proportion of children who use at least one information technology product for their own use is 63.8%. Other studies on the subject emphasize that digital addiction and its subtypes lead to many negative biopsychosocial consequences on adolescent health, such as vision loss, obesity, sleep disorders, anxiety, depression, and poor communication skills. Furthermore, existing literature highlights a significant relationship between digital addiction and cyberbullying. These data demonstrate that digital devices are an indispensable part of daily life among adolescents, and digital addiction should be considered a significant risk factor threatening adolescent mental health. Therefore, nursing approaches to combating digital addiction specific to adolescence are of great importance in terms of instilling healthy digital habits and creating a safe environment in the digital world. Approaches such as psychoeducation and cognitive behavioral therapy have been primarily preferred in combating digital addiction. In fact, studies on the subject frequently use terms such as problematic internet use or internet or technology addiction instead of digital addiction. However, these traditional approaches may be insufficient to achieve behavioral change in individuals. Therefore, there is a need to investigate the effectiveness of arts-based nursing interventions that incorporate more holistic, expressive, and creative processes for digital addiction, which is considered a multifaceted problem. At this point, art therapy offers the opportunity to reveal emotions, explore the inner world, and increase self-efficacy without the need for verbal expression. It is anticipated that art therapy can contribute to the development of healthy digital habits by reducing excessive use of digital technology in adolescents and can be an alternative area of interest for a more productive use of free time. A review of national and international literature reveals that art therapy or art-based approaches applied to adolescents: Although positive effects have been observed on psychological problems such as stress, anxiety, depression, internet, smartphone or game addiction, no studies have been found on how it can have a direct effect on digital addiction. Also, see. Digital addiction, like other types of addiction, cannot be resolved with a "zero use" approach; in this increasingly digital world, completely removing adolescents from technological devices is both impossible and detaches them from the demands of the age. Based on this, we believe that supporting adolescents' healthy use of digital devices should be the primary goal. In this context, this original research aims to fill the gap in the literature by examining the effects of an arts-based nursing intervention that helps develop healthy digital habits on digital addiction, cyberbullying, and self-efficacy in adolescents. Based on the findings of this study, it is anticipated that individual self-efficacy can be strengthened through arts-based approaches in combating digital addiction, a new generation of behavioral addictions. Furthermore, arts-based interventions are expected to provide a scientific basis for school health services, adolescent mental health programs, and nursing practices.

ELIGIBILITY:
Inclusion Criteria:

* Being a 6th-grade middle school student,
* The student and their parent must provide written consent to participate in the study,
* Understanding and speaking Turkish at a level sufficient to complete the data forms and participate in the sessions.

Exclusion Criteria:

* Having participated in a similar program within the last 6 months,
* Having a serious psychiatric diagnosis or physical disability that prevents participation in art activities.
* Not attending any two sessions,
* Requesting to leave the sessions,

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Digital Addiction Level | Baseline (Week 0) and immediately after the 8-week intervention
  Digital addiction will be measured using the 25-item self-report Digital Addiction Scale for Children, adapted into Turkish. It evaluates interpersonal relationships and internalized factors using a 5-point Likert scale, with total scores ranging from 25 to 125. Higher scores indicate a higher risk of digital addiction.
Cyberbullying and Victimization Levels | Baseline (Week 0) and immediately after the 8-week intervention
  Cyberbullying perpetration and victimization will be assessed using the Revised Cyberbullying Inventory-II (RCBI-II). The tool consists of 20 items across two parallel forms (perpetrator and victim), using a 4-point Likert scale, with total scores ranging from 1 to 80. Higher scores indicate higher levels of cyberbullying behaviors or victimization.
Self-Efficacy Level | Baseline (Week 0) and immediately after the 8-week intervention
  Self-efficacy will be measured using the 21-item Self-Efficacy Scale for Children. It consists of three subscales: academic, social, and emotional self-efficacy, with total scores ranging from 21 to 105. Higher scores indicate higher levels of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Koçak Uyaroğlu, Associate Professor, Study Director — Selcuk University; Esra Ünal, Research Assistant, Principal Investigator — Selcuk University

IPD SHARING:
Plan to Share IPD: No
IPD Sharing Plan:
  No
  IPD Sharing Description:
  Individual participant data (IPD) will not be shared due to ethical concerns and the involvement of a vulnerable population (adolescents). The study does not include prior consent for data sharing beyond the primary research team.
  IPD Sharing Access Criteria:
  Not applicable.

REFERENCES:
- [Background] Schulz van Endert T. Addictive use of digital devices in young children: Associations with delay discounting, self-control and academic performance. PLoS One. 2021 Jun 22;16(6):e0253058. doi: 10.1371/journal.pone.0253058. eCollection 2021. PMID 34157026
- [Background] Aziz N, Nordin MJ, Abdulkadir SJ, Salih MMM. Digital addiction: systematic review of computer game addiction impact on adolescent physical health. Electronics. 2021; 10(9): 996. doi:10.3390/electronics10090996
- [Background] Gorowska M, Tokarska K, Zhou X, Gola MK, Li Y. Novel approaches for treating Internet Gaming Disorder: A review of technology-based interventions. Compr Psychiatry. 2022 May;115:152312. doi: 10.1016/j.comppsych.2022.152312. Epub 2022 Apr 3. PMID 35405548
- [Background] Zhang B, Wang J, Abdullah AB. The effects of art therapy interventions on anxiety in children and adolescents: A meta-analysis. Clinics (Sao Paulo). 2024 Jun 26;79:100404. doi: 10.1016/j.clinsp.2024.100404. eCollection 2024. PMID 38936289
- [Background] Blomdahl C, Goulias A. Art therapy for adolescents with depression: feasibility and acceptability study in child and adolescent psychiatry. Art Therapy. 2025; 42(1): 14-23.
- [Background] Mittal S, Mahapatra M, Ansari SA. Effect of art therapy on adolescents' mental health. Российский Психологический Журнал. 2022; 19(4): 71-79.
- [Background] Hylton E, Malley A, Ironson G. Improvements in adolescent mental health and positive affect using creative arts therapy after a school shooting: a pilot study. The Arts in Psychotherapy. 2019; 65: 101586.
- [Background] Yanık D, Arslan R. Efficacy of technology addiction awareness training given to high school students: randomized controlled experimental study. OPUS Journal of Society Research. 2023; 20(54): 518-528.
- [Background] Uysal G, Balci S. Evaluation of a School-Based Program for Internet Addiction of Adolescents in Turkey. J Addict Nurs. 2018 Jan/Mar;29(1):43-49. doi: 10.1097/JAN.0000000000000211. PMID 29505460
- [Background] Agbaria Q. Cognitive behavioral intervention in dealing with Internet addiction among Arab teenagers in Israel. Int J Ment Health Addict. 2022 Jan 20:1-15. doi: 10.1007/s11469-021-00733-6. Online ahead of print. PMID 35075353
- [Background] Ime Y, Akyıl Y, Caglar A. The examination of the relationships among digital addiction, loneliness, shyness, and social anxiety in adolescents. Anales de Psicología/Annals of Psychology. 2024; 40(2): 236-241.
- [Background] Cimke S, Gurkan DY, Sirganci G. Determination of the psychometric properties of the digital addiction scale for children. J Pediatr Nurs. 2023 Jul-Aug;71:1-5. doi: 10.1016/j.pedn.2023.03.004. Epub 2023 Mar 20. PMID 36947896
- [Background] Meng SQ, Cheng JL, Li YY, Yang XQ, Zheng JW, Chang XW, Shi Y, Chen Y, Lu L, Sun Y, Bao YP, Shi J. Global prevalence of digital addiction in general population: A systematic review and meta-analysis. Clin Psychol Rev. 2022 Mar;92:102128. doi: 10.1016/j.cpr.2022.102128. Epub 2022 Jan 25. PMID 35150965
- [Background] Karabulut A. The effect of addiction education on digital addiction levels of university students. Journal of Medical Social Work. 2023; 21: 1-25.
- [Result] Bagatarhan T, Siyez DM. The digital addiction scale for children: psychometric properties of the Turkish version. Curr Psychol. 2023 Apr 22:1-11. doi: 10.1007/s12144-023-04675-1. Online ahead of print. PMID 37359651
- [Result] Topcu Ç, Erdur-Baker Ö. RCBI-II: The second revision of the revised cyber bullying inventory. Measurement and Evaluation in Counseling and Development. 2018; 51(1): 32-41.
- [Result] Hawi NS, Samaha M, Griffiths MD. The Digital Addiction Scale for Children: Development and Validation. Cyberpsychol Behav Soc Netw. 2019 Dec;22(12):771-778. doi: 10.1089/cyber.2019.0132. Epub 2019 Nov 22. PMID 31755742
- See also: Turkish Statistical Institute. (2024). Survey on information and communication technology usage in children. Retrieved April 29, 2025. — https://data.tuik.gov.tr/Bulten/Index?p=Cocuklarda-Bilisim-Teknolojileri-Kullanim-Arastirmasi-2024-53638